CLINICAL TRIAL: NCT04435054
Title: Screening for NAFLD-related Advanced Fibrosis in High Risk popuLation: Optimization of the Diabetology Pathway Referral Using Combinations of Non-invAsive Biological and elastogRaphy paramEters
Brief Title: Screening for NAFLD-related Advanced Fibrosis in High Risk Population in Diabetology.
Acronym: NAFLD-CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 69HCL20_0033
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: NAFLD; Type 2 diabete; Obesity; Advanced fibrosis; Cirrhosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Obesity; Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non invasive tests (Other)
  Interventions: Diagnostic Test: Non-invasive blood-based and imaging-based tests for the screening of NAFLD-related advanced fibrosis.

INTERVENTIONS:
Diagnostic Test: Non-invasive blood-based and imaging-based tests for the screening of NAFLD-related advanced fibrosis. — Non-invasive blood biological tests - NAFLD Fibrosis Score, FIB-4, Fibrotest, FibrometerNAFLD
  Non-invasive imaging:
  - Transient elastography (FibroScan), Shear Wave imaging, Magnetic resonance imaging (MRI-PDFF and MRE) in a subgroup of participants.

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) is being recognized as one of the most prevalent causes of chronic liver disease worldwide. The current strategy proposed by the EASL/EASO/EASD European guidelines for the screening of nonalcoholic fatty liver disease (NAFLD) in high-risk population such as type 2 diabetes and patients with obesity leads to an over-referral in hepatology clinics. The proposed study will investigate the optimal strategy for the screening of NAFLD-related advanced fibrosis in patients at high risk of fibrotic NAFLD, such as patients with T2DM or obesity by maximizing the positive predictive value (PPV) using non-invasive blood and elastography-based biomarkers in endocrinology/diabetology clinics in order to reduce the over-referral to hepatology clinics.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged between 40 and 80 years old,
* Patients with diagnosis of T2DM* or obesity (defined according to World Health Organization as a BMI≥ 30 kg/m2)
* Patient with hepatic steatosis determined by conventional abdominal ultrasound as defined by the EASL/EASO/EASD European guidelines.
* Patient who agrees to be included in the study and who signs the informed consent form,
* Patient affiliated to a healthcare insurance plan.

Exclusion Criteria:

* Evidence of other causes of chronic liver disease:
* History of ingestion of medications known to produce steatosis in the previous 6 months.
* Evidence of cirrhosis or previously known cirrhosis based on the results from previous liver biopsy or history of portal hypertension presented by ascites, hepatic encephalopathy or varices
* Presence of regular and/or excessive use of alcohol (defined as >30g/day for males and >15g/day for females) for a period longer than 2 years at any times in the last 10 years
* The subject is a pregnant or nursing female
* Life expectancy less than 5 years
* History of known HIV infection
* History of type 1 diabete
* BMI ≥ 40 kg/m2
* Mentally unbalanced patients, under supervision or guardianship,
* Patient deprived of liberty,
* Patient who does not understand French/ is unable to give consent,
* Patient already included in a trial who may interfere with the study or in a period of exclusion following participation in a previous study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2023-10-28 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Presence of individual F0 to F4 stage of fibrosis | 6 months
  The presence of individual F0 to F4 stage of fibrosis as defined by histological stage in the liver biopsy using the NASH CRN Scoring System.

SECONDARY OUTCOMES:
Fibroscan | 6 months
  The presence of liver stiffness measured using Fibroscan (VCTE) ≥ 7 kPa.

CONTACTS AND LOCATIONS:
Overall Officials: Cyrielle CAUSSY, MD, Principal Investigator — Hospices Civils de Lyon
Locations (3):
- France (3):
  - Centre Hospitalier Universitaire Dijon Bourgogne, Dijon
  - CHU de Nantes, Nantes
  - Hôpital Lyon Sud, Pierre-Bénite

REFERENCES:
- [Result] Caussy C, Verges B, Leleu D, Duvillard L, Subtil F, Abichou-Klich A, Hervieu V, Milot L, Segrestin B, Bin S, Rouland A, Delaunay D, Morcel P, Hadjadj S, Primot C, Petit JM, Charriere S, Moulin P, Levrero M, Cariou B, Disse E. Screening for Metabolic Dysfunction-Associated Steatotic Liver Disease-Related Advanced Fibrosis in Diabetology: A Prospective Multicenter Study. Diabetes Care. 2025 Jun 1;48(6):877-886. doi: 10.2337/dc24-2075. PMID 39887699